CLINICAL TRIAL: NCT01233973
Title: Using Videos to Improve Understanding of the Delivery of End-of-life Medical Care in Non-hospital Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Faculty, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010-P-000180
Record Dates: First submitted 2010-11-01; First posted 2010-11-04 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Elderly
Keywords: nursing home; advance care planning
MeSH Terms: interventions — Decision Support Techniques; Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control subjects (No Intervention): verbal narrative of advance care planning
- intervention group (Experimental): video decision aid viewed by subjects
  Interventions: Other: video decision aid

INTERVENTIONS:
Other: video decision aid — video
  Other Names: decision aid; film
  Arms: intervention group

SUMMARY:
To compare the decision making of elderly subjects having a verbal advance care planning discussion compared to subjects using a video.

DETAILED DESCRIPTION:
A.1. Aim 1: To recruit 101 subjects over the age of 64 who are newly admitted to a nursing home facility and randomly assign these subjects to one of two advance care planning (ACP) modalities: 1. a video visually depicting the Goals of Care (Life Prolonging Care, Limited Care, and Comfort Care) (intervention) or 2. a verbal narrative describing the Goals of Care (control) encountered if the subject becomes very ill.

Hypothesis 1: It is feasible to recruit and randomize newly admitted elderly subjects to each of the ACP modalities.

A.2. Aim 2: To compare the care preferences for their primary goal of care (i.e., life-prolonging care, limited care, or comfort care) among 101 subjects randomized to video vs. verbal narrative intervention for ACP.

Hypothesis 2: Subjects randomized to the video intervention will be significantly more likely to opt for comfort care (vs. life-prolonging or limited care) as the primary goal of care compared to those randomized to the verbal narrative.

A.3. Aim 3: To compare knowledge assessment of the Goals of Care of 101 subjects randomized to video vs. verbal narrative intervention for ACP.

Hypothesis 3: When compared to subjects randomized to the verbal narrative arm, subjects in the video group will have higher knowledge assessment scores when asked questions regarding their understanding of the Goals of Care.

ELIGIBILITY:
Inclusion Criteria:

* over age of 64
* have decision making capacity

Exclusion Criteria:

* do not speak English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
preference for medical care | 5 minutes after the survey
  preference for care at the end of life

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Volandes, Principal Investigator — MGH
Locations (1):
- MGH, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Volandes AE, Brandeis GH, Davis AD, Paasche-Orlow MK, Gillick MR, Chang Y, Walker-Corkery ES, Mann E, Mitchell SL. A randomized controlled trial of a goals-of-care video for elderly patients admitted to skilled nursing facilities. J Palliat Med. 2012 Jul;15(7):805-11. doi: 10.1089/jpm.2011.0505. Epub 2012 May 4. PMID 22559905